CLINICAL TRIAL: NCT01737411
Title: Surgical vs. Medical Treatment of Urge Urinary Incontinence in Women
Acronym: URGE-I
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Klinikum der Universität Köln (Other)
Responsible Party: Principal Investigator, Professor Dr. Wolfram Jäger, Professor, Klinikum der Universität Köln
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: URGE-I; URGE-I (Other: OB/GYN); URGE-I (Other: OB/GYN Köln); 11-016 (Other: University of Köln)
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Urge Urinary Incontinence
Keywords: surgery, solifenacin, urge urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Urge | interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- solifenacin (Active Comparator): 10 mg solifenacin per day for three months
  Interventions: Drug: solifenacin
- cesa/vasa (Experimental): repair of USL
  Interventions: Procedure: cesa/vasa

INTERVENTIONS:
Drug: solifenacin
  Other Names: VESICUR
  Arms: solifenacin
Procedure: cesa/vasa — surgical repair of USL
  Arms: cesa/vasa

SUMMARY:
The purpose of this study is to determine if pelvic surgery can improve urge urinary incontinence in women more than standard medical treatment.

DETAILED DESCRIPTION:
Urge Urinary Incontinence affects 30% of postmenopausal women. The etiology is unknown therefore treatment is symptomatic. For that purpose the nerval stimulation of the bladder muscle is interfered by several drugs, e.g. solifenacin.

We observed that the surgical repair of critical pelvic structures, i.e. the uteri-sacral ligaments (USL) can restore continence in a considerable number of patients.

In this study the surgical treatment is compared with the solifenacin treatment. According to outcome after three months patients who are still incontinent are referred to the opposite treatment group.

Outcome will be differentiated in cure (primary aim) and improvement of symptoms (secondary aim).

ELIGIBILITY:
Inclusion Criteria:

* urge urinary incontinence

Exclusion Criteria:

* stress urinary incontinence
* cancer disease of the females genital tract
* pregnancy
* neurologic/psychological reasons for incontinence
* body weight >100kg
* previous urogynecological surgery (TVT)
* syndrome of dry overactive bladder (>20 micturitions within 24 hours)

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
cure from urge urinary symptoms | 12 months
  At the start of the study urge symptoms are categorized from 0 (no symptom for the specific item) to 2 (worst expression of symptom). Cure is defined when sum of category points is 0, improvement is defined when category points are less after than before treatment

SECONDARY OUTCOMES:
cure from urge urinary symptoms | 12 months
  When the assigned first line treatment did not cure patients receive the treatment of the other arm (cross-over). Before cross-over urge symptoms of each patient are categorized from 0 (no symptom for the specific item) to 2 (worst expression of symptom). Cure is defined when sum of category points is 0, improvement is defined when category points are less after than before treatment

OTHER OUTCOMES:
stress incontinence | 12 months
  Some patients develop a stress incontinence after surgical treatment. That is controlled by provocation tests.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfram H Jager, PhD, Study Director — Study Supervisor
Locations (1):
- Abt. Beckenbodenchirugie der Universitäts-Frauenklinik Köln, Cologne, North Rhine-Westphalia, Germany